CLINICAL TRIAL: NCT04603989
Title: A Randomized, Double-blind, Placebo-controlled, Sequential Parallel Group, Multiple Ascending Doses Study Following Intravenous Administration in Healthy Chinese Volunteers to Evaluate the Safety, Tolerability, and Pharmacokinetics of HNC042
Brief Title: A Study of HNC042 in Healthy Chinese Subjects to Evaluate the Safety, Tolerability, and Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Henovcom Bioscience Co. Ltd. (Industry)
Collaborators: Heilongjiang Zhenbaodao Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HNC042-102; ZBD1042-CSP01 (Other Grant/Funding Number: Heilongjiang Zhenbaodao Pharmaceutical Co., Ltd)
Record Dates: First submitted 2020-10-13; First posted 2020-10-27 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2020-08

CONDITIONS: Influenza
Keywords: Neuraminidase inhibitor
MeSH Terms: conditions — Influenza, Human | interventions — Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HNC042 (Experimental): HNC4042 for injection,freeze-dried powder,multiple ascending doses, Intravenous route
  Interventions: Drug: HNC042 for Injection
- Placebo (Placebo Comparator): Placebo, multiple ascending doses, Intravenous route
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: HNC042 for Injection — HNC042,freeze-dried powder,multiple ascending doses, Intravenous route Multiple doses, daily for 7 days, doses: 300mg to 1200mg
  Arms: HNC042
Drug: Placebo Comparator — Placebo , Intravenous route , multiple ascending doses
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety , tolerability and pharmacokinetics after multiple ascending of HNC042 given to healthy Chinese volunteers, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* volunteers can communicate well with the investigator, understand and comply with the relevant requirements of the study, understand and sign the informed consent
* Healthy adult male or female volunteers, age 18-65 years，
* BMI between 19-26 kg/m2,and male body weight not less than 50.0kg,female body weight not less than 45.0kg .
* volunteers with normal renal function

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Number of subjects with abnormal vital signs | Between screening and 15 days after the last dose
  To evaluate the safety and tolerability of HNC042 in comparison with placebo after multiple intravenous dose in healthy Chinese subjects in terms of abnormal vital signs
Number of subjects with abnormal laboratory | Between screening and 15 days after the last dose
  To evaluate the safety and tolerability of HNC042 in comparison with placebo after multiple intravenous dose in healthy Chinese subjects in terms of abnormal laboratory
Number of subjects with abnormal electrocardiogram | Between screening and 15 days after the last dose
  To evaluate the safety and tolerability of HNC042 in comparison with placebo after multiple intravenous dose in healthy Cjinese subjects in terms of abnormal electrocardiogram
Number of subjects with abnormal physical examination | Between screening and 15 days after the last dose
  To evaluate the safety and tolerability of HNC042 in comparison with placebo after multiple intravenous dose in healthy Cjinese subjects in terms of abnormal physical examination
Number of subjects with adverse reactions at injection site | Between screening and 15 days after the last dose
  To evaluate the safety and tolerability of HNC042 in comparison with placebo after multiple intravenous dose in healthy Cjinese subjects in terms of adverse reactions at injection site
Number of subjects with adverse events | Between screening and 15 days after the last dose
  To evaluate the safety and tolerability of HNC042 in comparison with placebo after multiple intravenous dose in healthy Cjinese subjects in terms of adverse events
Number of subjects with clinical symptoms | Between screening and 15 days after the last dose
  To evaluate the safety and tolerability of HNC042 in comparison with placebo after multiple intravenous dose in healthy Cjinese subjects in terms of clinical symptoms

SECONDARY OUTCOMES:
Pharmacokinetics of HNC042 in plasma: Cmax | Between Day 1 to 7 days
  To characterize the pharmacokinetic parameters：Cmax of HNC042 after the the first day administer .
Pharmacokinetics of HNC042 in plasma: Tmax | Between Day 1 to 7 days
  To characterize the pharmacokinetic parameters：Tmax of HNC042 after the the first day administer .
Pharmacokinetics of HNC042 in plasma: AUC0-last | Between Day 1 to 7 days
  To characterize the pharmacokinetic parameters：AUC0-last of HNC042 after the the first day administer .
Pharmacokinetics of HNC042 in plasma: AUC0-∞ | Between Day 1 to 7 days
  To characterize the pharmacokinetic parameters： AUC0-∞ of HNC042 after the the first day administer .
Pharmacokinetics of HNC042 in plasma:t1/2 | Between Day 1 to 7 days
  To characterize the pharmacokinetic parameters： t1/2 of HNC042 after the the first day administer .
Pharmacokinetics of HNC042 in plasma:MRT | Between Day 1 to 7 days
  To characterize the pharmacokinetic parameters： MRT of HNC042 after the the first day administer .
Pharmacokinetics of HNC042 in plasma:CL | Between Day 1 to 7 days
  To characterize the pharmacokinetic parameters：CL of HNC042 after the the first day administer .
Pharmacokinetics of HNC042 in plasma:Vd | Between Day 1 to 7 days
  To characterize the pharmacokinetic parameters：Vd of HNC042 after the the first day administer .

CONTACTS AND LOCATIONS:
Overall Officials: Lu Xiang, MD, Principal Investigator — Nanjing Medical University
Locations (1):
- Jiang Yuting, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No